CLINICAL TRIAL: NCT05103670
Title: Ventilation/Perfusion PET/CT With Galligas and 68Ga-MAA for Regional Lung Function Assessment After Pulmonary Embolism
Acronym: EOLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC21.0139 (EOLE)
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Embolism; Dyspnea
Keywords: Ventilation/perfusion PET/CT; Galligas; 68Ga-MAA
MeSH Terms: conditions — Pulmonary Embolism; Dyspnea; Respiratory Aspiration | interventions — Ventilation

STUDY DESIGN:
Intervention Model Description: EOLE is an ancillary study which selects patients included in the RAMBO study. The RAMBO study is a 2-arm-parallel study which patients included in one arm will undergo a 3-month pulmonary rehabilitation, and the patients included in the other arm won't. The EOLE study will include patients in both arms of the RAMBO study. All participants will undergo a PET/CT scan at inclusion and at 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients undergoing a Ventilation/Perfusion PET/CT at inclusion and 3 months later (Experimental): EOLE is an ancillary study which selects patients included in the RAMBO study. The RAMBO study is a 2-arm-parallel study which patients included in one arm will undergo a 3-month pulmonary rehabilitation, and the patients included in the other arm won't. The EOLE study will include specific patients in both arms of the RAMBO study, and all of the participants will undergo a PET/CT scan at the inclusion and 3 months later.
  Interventions: Procedure: Ventilation/Perfusion PET/CT with Galligas and 68Ga-MAA

INTERVENTIONS:
Procedure: Ventilation/Perfusion PET/CT with Galligas and 68Ga-MAA — 32 patients will undergo a Ventilation/Perfusion PET/CT with Galligas and 68Ga-MAA at the inclusion and 3 months later.

SUMMARY:
In patients with pulmonary embolism (PE), after three or six months of anticoagulation, persistent dyspnea and impairment of quality of life are observed in at least 30% of cases.

The "RAMBO" trial is a French academic, multicenter, randomized (1:1 ratio), parallel arm, controlled, that aimed to assess the efficacy of pulmonary rehabilitation (PR) on the quality of life in patients with an acute symptomatic PE treated with anticoagulant therapy during at least 3 months and who present an impairment of quality of life and/or persistent dyspnea despite anticoagulant therapy.

Ventilation/Perfusion (V/Q) PET/CT is a novel imaging modality for the assessment of regional lung function. The same carrier molecules as conventional V/Q imaging are used, but they are labeled with 68Gallium, a ß+ isotope, instead of 99mTc, allowing acquisition of images with PET technology.

The EOLE study is an ancillary pilot study of the RAMBO trial, in which patients will benefit, in addition to the extensive work up scheduled as per study protocol, from a V/Q PET/CT scan before and after PR. The aim of the study is to assess the impact of PR on regional lung function with lung V/Q PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in the RAMBO study, whose inclusion criteria are: Age ≥ 18 years; Patient treated with at least 3 months and up to 8 months of anticoagulation for an acute symptomatic PE diagnosed according the ESC and ACCP guidelines; Patients who have a PembQol score ≥ 10% and whose total scores for the subgroups Q1 (dyspnea) and Q4 (impact of daily life) are ≥ 10%.
* Patients planned to be randomized
* Abnormal conventional V/Q scan at V1
* Give consent to participate to the EOLE study

Exclusion Criteria:

* Non inclusion criteria of the RAMBO trial:
* Previsible inability to perform the effort test and/or PR
* Presence of CTEPH according to international guidelines
* Patients treated for acute PE with anticoagulants for more than 8 months
* Active cancer or in remission for less than two years
* Dyspnea post - COVID due to parenchymal injuries
* Post-COVID hyperventilation syndrome without pulmonary vascular perfusion sequelae
* Physical or psychological inability to undertake PR
* Isolated or more distal segmental PE
* Neuro-muscular disease with PR contraindication.
* Cardiac insufficiency (unstable coronary artery disease)
* Severe respiratory failure (long-term oxygen therapy, pulmonary hypertension)
* Chronic dyspnea MMRC ≥ 2 before PE
* Cardiac or respiratory rehabilitation in the previous year
* Indication to urgent PR within 6 months at the time of inclusion
* Life expectancy of less than 12 months
* Inability to give consent
* Patient under guardianship or curatorship
* Patient deprived of liberty by an administrative or judicial decision
* Patient has not social security affiliation or who don't beneficiary of such social security

After initial PR work up, patients with following criteria cannot be included:

* Incapacity to perform the effort test
* Effort test stopped because of hemodynamic intolerance
* Cardiac failure discovered after PR work up

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular obstruction index (PVOI) on V/Q PET/CT imaging. | 3 months
  Expressed as a percentage of whole lung

SECONDARY OUTCOMES:
Pulmonary ventilation impairment index on V/Q PET/CT imaging. | 3 months
  Expressed as a percentage of whole lung

CONTACTS AND LOCATIONS:
Locations (1):
- LEROUX Pierre-Yves, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.